CLINICAL TRIAL: NCT03065049
Title: Peer-Facilitated Physical Activity Intervention Delivered During Methadone Maintenance
Brief Title: Transforming Recovery Through Exercise and Community
Acronym: TREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1609-001; 1R21DA041553-01A1 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-02-27 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Opioid-use Disorder
Keywords: Physical Activity; Peer-facilitation; Methadone Maintenance Therapy
MeSH Terms: conditions — Opioid-Related Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer-PA+Fitbit (Experimental): Participants will engage in a 12-week physical activity intervention guided by a peer-facilitator at the methadone clinic they receive treatment. Participants will attend weekly groups, engage in a guided walking group, and utilize the Fitbit to self-monitor physical activity.
  Interventions: Behavioral: Peer-Facilitated Counseling; Behavioral: Fitbit activity tracker
- Fitbit Only (Active Comparator): Participants will be given a Fitbit activity tracker along with brief advice for increasing physical activity.
  Interventions: Behavioral: Fitbit activity tracker
- Usual Care (No Intervention): Participants do not receive any intervention but participate in the assessments only.

INTERVENTIONS:
Behavioral: Peer-Facilitated Counseling — Participants will engage in a 12-week physical activity intervention guided by a peer-facilitator at the methadone clinic they receive treatment. Participants will attend weekly groups, engage in a guided walking group, and utilize the Fitbit to self-monitor physical activity.
  Arms: Peer-PA+Fitbit
Behavioral: Fitbit activity tracker — Participants will be given a Fitbit activity tracker to monitor physical activity.
  Arms: Fitbit Only; Peer-PA+Fitbit

SUMMARY:
The primary aim of this study is to develop a feasible, acceptable, and effective multilevel physical activity (PA) intervention that addresses both individual and interpersonal factors that can be easily scalable and delivered in the context of a methadone clinic. To do so, the investigators will train methadone maintenance treatment (MMT) patients who are already engaging in PA at public health recommended levels to deliver a group-based PA intervention to physically inactive MMT patients at a large community-based methadone clinic. Through the development of interpersonal relationships and social support, the investigators expect that MMT peers who have successfully navigated challenges associated with PA in this population (i.e. depression, smoking, triggers for drug use in environment) will help physically inactive MMT patients increase self-efficacy and motivation for initiating and sustaining PA.

DETAILED DESCRIPTION:
Opioid Use Disorders (OUDs) are a highly prevalent and costly public health concern in the United States, with over 2.59 million Americans qualifying for abuse or dependence of opioids in 2015. Methadone maintenance treatment (MMT), involving daily distribution of methadone at regulated clinics, is the most common treatment for opioid use disorder. While MMT has been effective in helping OUD patients improve their quality of life, the overwhelming majority of these patients continue to engage in unhealthy lifestyles (e.g., physical inactivity and cigarette smoking) that lead to significant physical and mental health morbidities. For example, patients in MMT have much higher rates of cardiovascular disease, diabetes, hypertension, obesity, depression, sleep difficulties, and cognitive impairments than age-matched controls, which lead to premature death. Given the mental health, physical health, and drug use related benefits of physical activity (PA), interventions targeting increases in PA in patients receiving MMT could have a significant impact on reducing their overall morbidity and mortality.

To date, few PA studies have been conducted with substance abusing populations - and, only one small pilot study with MMT patients. The goal of this project is to develop a feasible, acceptable and effective multilevel PA intervention that addresses both individual and interpersonal factors that can be easily scalable and delivered in the context of a health care setting (i.e., methadone clinics). To do so, the investigators are proposing to train MMT patients who are already engaging in PA at public health recommended levels to deliver a group-based PA intervention to physically inactive MMT patients at SSTAR Lifeline, a large community-based methadone clinic in Fall River, Massachusetts. Peer-facilitated interventions for self-management skills are common in the care of patients with chronic medical conditions. Peers may play a particularly important role in increasing physical activity in MMT, as this population faces unique and significant barriers to PA (e.g., depression, smoking, minimal social supports). Through the development of interpersonal relationships, the investigators expect that MMT peers who have successfully navigated these challenges will help physically inactive MMT patients increase self-efficacy and motivation for initiating and sustaining PA.

The aims of the study include:

1. PHASE 1 (Peer-PA Manual Development):

   * To develop a theoretically-informed peer-facilitated PA plus Fitbit (Peer-PA+Fitbit) intervention specific to SSTAR Lifeline, in order to help patients in MMT increase levels of physical activity.

     1. Focus groups will be conducted with: 1) MMT patients who are currently physically active and 2) MMT patients who are NOT meeting recommended PA levels to help inform intervention development.
     2. The investigators will: (1) develop a manualized Peer-PA intervention (that includes the use of a Fitbit activity monitor for self-monitoring PA and additional social networking), (2) create a training protocol for MMT patients to become peer-facilitators, and (3) identify safe, walkable paths in participant neighborhoods.
2. PHASE 2 (Open Pilot):

   * An open pilot trial will be conducted with 20 MMT patients to determine the feasibility, acceptability, and short term increases in PA of the Peer-PA+Fitbit intervention. At the end of 3 months:

     1. Feedback will be obtained on Peer-PA+Fitbit from both the MMT peers and participants through self-report measures and qualitative interviews.
     2. Adherence to the intervention will be determined through group attendance and Fitbit data.
     3. Short-term increases in physical activity levels will be examined through objectively measured PA.
3. PHASE 3 (Randomized Clinical Trial; RCT)

To conduct a 3-arm preliminary RCT of Peer-PA+Fitbit compared to Fitbit Only and compared to Usual Care (UC) among 150 MMT patients. We hypothesize that, Peer-PA+Fitbit will be superior to Fitbit Only and that Fitbit Only will be superior to UC on the following:

1. Higher levels of short-term (3-month) and long-term (6- and 12-month) objectively-measured steps/day and moderate-to-vigorous physical activity (MVPA)
2. Fewer days of drug use and lower levels of depression and anxiety symptoms at each follow-up
3. Higher levels of theoretically-relevant, PA-related variables including: self-efficacy, internal motivation, and social support at 3- and 6-month follow-ups

ELIGIBILITY:
Inclusion Criteria:

* receiving MMT at SSTAR and planning to remain in treatment for the next 6 months
* low active (i.e., less than 90 minutes of MIPA per week for the past 6 months)
* has access to a computer connected to the internet or a smartphone compatible with the Fitbit application

Exclusion Criteria:

* a history of psychotic disorder or current psychotic symptoms
* current suicidality or homicidality
* marked organic impairment according to responses to the diagnostic assessments
* physical or medical problems that would not allow safe participation in a program of moderate intensity physical activity (i.e., not medically cleared by methadone clinic physician)
* current pregnancy or intent to become pregnant during the next 12 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate-to-vigorous physical activity (MVPA)/week | 12 month
  Measured by accelerometry

SECONDARY OUTCOMES:
Acceptability of the Intervention assessed with the Client Satisfaction Questionnaire | 12 weeks
  Client Satisfaction Questionnaire (CSQ-8)
  * Total score = summation of scores from each question
  * Maximum score for each question is 4 points (range from 1 - 4)
  * Maximum score for the measure is 32
  * The higher the total score, the better the acceptability
level of depressive symptoms | 12 month
  Center for Epidemiological Studies Depression Scale (CES-D)
  * Total score = summation of scores from each question
  * Scoring: 0 = Rarely or None of the time (Less than 1 day), 1 = Some or a Little of the time (1-2 days), 2 = Occasionally or a Moderate Amount of time (3-4 days), 3 = Most or All of the time (5-7 days)
  * Maximum score for the measure is 60
  * Higher scores = higher symptoms of depressive symptomatology
level of anxiety symptoms | 12 month
  Generalized Anxiety Disorder 7-item scale (GAD-7)
  * Total score = summation of scores from each question
  * Scoring for items #1-7: 0 = Not at all, 1 = Several days, 2 = Over half the days, 3 = Nearly every day
  * Item #8 is qualitative (not scored) and has the following answer choices: Not difficult at all, Somewhat difficult, Very difficult, Extremely difficult
  * Maximum score for the measure is 21
  * Higher scores = higher anxiety severity

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Abrantes, Ph.D., Principal Investigator — Butler Hospital; Michael Stein, M.D., Principal Investigator — Boston University
Locations (1):
- Stanley Street Treatment and Resources (SSTAR) Lifeline, Fall River, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided